CLINICAL TRIAL: NCT04073628
Title: The Long-term Impact of a Light Intervention on Sleep Physiology and Cognition in Mild Cognitive Impairment
Brief Title: The Long-term Impact of a Light Intervention on Sleep and Cognition in Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Rutgers University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mariana Figueiro, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 21-0019; R01AG062288 (NIH)
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
Keywords: Mild Cognitive Impairment, sleep and memory
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: In a single-arm, randomized, placebo-controlled (non-active comparison lighting intervention), between-subjects study, we will investigate the effect of long-term exposure (6 months) to a lighting intervention, which is designed to promote circadian entrainment.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Lighting intervention (Active Comparator): The active lighting intervention will provide high circadian stimulation during the day produced by light sources that provide moderate light levels of spectra that are tuned to the sensitivity of the circadian system. Combining spectrum and light level, the intervention will allow us to: (1) use a light source that will stimulate the circadian system and (2) provide the participants with options as to how the light treatment will be delivered
  Interventions: Device: Lighting Intervention
- Control Lighting Intervention (Placebo Comparator): The control lighting intervention will consist of low levels of a warm light source designed not to impact the circadian system.
  Interventions: Device: Lighting Intervention

INTERVENTIONS:
Device: Lighting Intervention — Lighting Intervention consisting of a cool or warm light source.

SUMMARY:
To investigate the impact of a long-term light treatment intervention on sleep physiology and memory in mild cognitively impaired and mild Alzheimer's disease patients living at home. The goal is also to measure the impact of the lighting intervention on caregivers' sleep, cognition, depression, and quality of life.

DETAILED DESCRIPTION:
The current application proposes to investigate the impact of a long-term light treatment intervention on sleep physiology and sleep-dependent cognitive processes in mild cognitive impairment (MCI) and mild Alzheimer's disease (AD) patients. The premise is that older adults, especially those with cognitive impairment, are often in continuous dim light, which leads to circadian misalignment. Circadian misalignment impacts the close relationship between homeostatic and circadian processes, which can reduce memory-related sleep features. The hypothesis is that a lighting intervention technology (LIT), designed to promote circadian entrainment, will improve sleep by aligning the two sleep processes (circadian and homeostatic) and, thus improve cognition. In addition to improving patients' lives, LIT has the potential to reduce the overnight burden on caregivers. Thus, an exploratory goal is to also measure the impact of LIT on caregivers' sleep, cognition, depression, and quality of life.

ELIGIBILITY:
Inclusion Criteria for MCI/Mild AD Participant:

* Subject has diagnosis of amnestic mild cognitive impairment (MCI) or mild Alzheimer's disease (AD), as defined by a Montreal Cognitive Assessment (MoCA) score between 17 and 24 and those who fall between 0.5-4.0 and 4.5-9.0 in the Clinical Dementia Rating Scale Sum of Boxes (CDR-SOB) instrument
* Subject has sleep disturbance indicated by a score >5 on the Pittsburgh Sleep Quality Index and sleep efficiency below 80% as indicated via actigraphy
* Subject resides in his/her home, independent living, or assisted living facilities with a caregiver.

Exclusion Criteria for MCI/Mild AD Participant:

* Subject diagnosed with another brain disease that fully explains the dementia (extensive brain vascular disease, Parkinson's disease, dementia with Lewy bodies, traumatic brain injury, or multiple sclerosis)
* Subject resides in a skilled nursing facility or long-term care
* Subject has had recent changes in psychotropics (14 days)
* Subject has major organ failure (e.g., kidney failure)
* Subject has uncontrolled generalized disorders such as hypertension or diabetes
* Subject has obstructing cataracts, macular degeneration, and/or blindness
* Subject has undergone cataract surgery and received an intraocular lens coated with ultraviolet- and blue-blocking filters (400-440/440-500 nm)
* Subject diagnosed with severe sleep apnea; using the Sleep Apnea scale of the Sleep Disorders Questionnaire (SA-SDQ) the study will use a score of 29 as a cutoff for men and a cutoff of 26 for women
* Subject diagnosed with restless leg syndrome (RLS); using the International Restless Legs Scale (IRLS), the study will use a cutoff of ≥11 as a positive screen for RLS
* Subject has a history of severe photosensitivity dermatitis, severe progressive retinal disease (e.g., macular degeneration), or a permanently dilated pupil (e.g., after certain types of cataract surgery)

For caregivers, we will accept those who:

* Live with the patients
* Are not diagnosed with dementia (MOCA between 25 and 30 and CDR=0)
* Understand English
* Are willing to help with the study
* No other inclusion/exclusion criteria will be used for enrolling caregivers. There is no age requirement for caregivers.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Cognition using the Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog) | Will be administered at baseline and the end of weeks 9, 17, 25 and 37
  Change in cognition of the MCI participant will be assessed utilizing the Alzheimer's Disease Assessment Scale-Cognitive to capture subtler changes in cognitive performance. The ADAS-Cog is the most widely used general cognitive measure in clinical trials of Alzheimer's disease. The ADAS-Cog assesses multiple cognitive domains including memory, language, praxis, and orientation.

SECONDARY OUTCOMES:
Depression using the Geriatric Depression Scale (GDS) | Will be administered at baseline and the end of weeks 9, 17, 25 and 37
  Change in depression of the MCI participant will be assessed via the Geriatric Depression Scale (GDS). The GDS is an instrument used to measure depression in healthy adults. We will use a short version of the GDS consisting of 15 questions. Ten of the questions indicate the presence of depression when answered positively, and the other five questions indicate depression when answered negatively. A lower score indicates less depressive symptoms.
Quality of Life using the Dementia Quality of Life Instrument (DQoL) | Will be administered at baseline and the end of weeks 9, 17, 25 and 37
  Change in quality of life of the MCI participant will be assessed with the Dementia Quality of Life Instrument (DQoL), via interview format. The DQoL measures self-esteem, positive affect/humor, negative affect, feelings of belonging, and sense of aesthetics. The DQoL consists of 29 items, grouped into five subscales according to domain. Subjects are instructed to answer using a 5-point response scale.
Light Exposure measurement in MCI Participants | Will be worn for seven days during baseline and seven days during weeks 9, 17, 25 and 37
  MCI participants will be given a daysimeter and asked to wear it as a pendant during all times while awake over the course of seven days during assessment weeks. The daysimeter will be used to monitor the total amount of circadian light received by the participant during the intervention weeks.
Sleep Efficiency in the MCI Participant | Will be worn for seven days during baseline and for seven days during weeks 9, 17, 25 and 37
  MCI participants will be asked to wear an actigraph for seven days during the assessment weeks. A positive change in sleep efficiency is better.
Cognition using the Montreal Cognitive Assessment (MoCA) tool | Will be administered at baseline and the end of weeks 9, 17, 25 and 37
  Change in cognition of the MCI participant will be assessed by utilization of the Montreal Cognitive Assessment (MoCA) tool. The MoCA is a one-page, 30-point test that can be administered in 10 minutes. It assesses short-term memory, visuospatial abilities, executive functions, attention, concentration and working memory, language, and orientation to time and place. In a validation study, it was shown to be a promising tool for detecting mild cognitive impairment and early Alzheimer's disease onset compared to the Mini Mental State Exam.
Cognition using the Word Pairs Associates (WPA) Task | Will be administered at baseline and the end of weeks 9, 17, 25 and 37
  Change in cognition of the MCI participant will be assessed by the Word Pairs Associate (WPA) task, in which subjects are visually presented with word-nonsense word pairs, to maximize the novel episodic and associative declarative memory demands of the task and minimize the semantic demands of the task. Participants are presented with 48 word-pairs in the evening WPA task session. Recognition tests are assessed both immediately following the encoding session, and delayed during retrieval (24 hours later to avoid circadian confounds). For the test, participants are presented with 40 intact word pairs (leaving off the first and last four pairs to avoid primacy and recency effects), as well as 40 rearranged word pairs (foils). Each word pair is displayed for 3000 milliseconds followed by a response prompt asking for a discrimination of whether the two words were shown together as a pair in the study list.
Sleep Quality in the MCI Participant using the Pittsburgh Sleep Quality Index (PSQI) | Will be administered at baseline and the end of weeks 9, 17, 25 and 37
  Change in sleep quality of the MCI participant will be assessed utilizing the Pittsburgh Sleep Quality Index (PSQI). The PSQI is composed of 19 items that generate seven component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction). The sum of the seven component scores yields a single global score. A global score >5 is considered to indicate sleep disturbances. A lower score indicates improvement in sleep quality.
Cognition using the Working Memory (WM) Task | Will be administered at baseline and the end of weeks 9,17, 25 and 37
  Change in cognition of the MCI participant will be assessed by the Working Memory (WM) task, comprised of nine practice and 20 test trials. Participants view a serial visual display of letters and math problems. They are asked to hold the letters in memory while simultaneously determining if the simple math problems are correct. Each of the simple math equation is on the screen for 3000 ms and each letter is presented for 1000 ms. Participants are instructed to press the "M" key with their right hand if the simple math equation is correct and press the "V" key with their left hand if the equation is not correct. Math performance is measured in percent correct. After each trial, a question mark appears on the screen to signal the response period. Participants are asked to enter the letters in the same order they were presented. Participants are tested in the WM task before a night of sleep and 24 hours later. Performance is assessed by calculating Accuracy and Reaction Time (RT).

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Figueiro, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, Albany, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No